CLINICAL TRIAL: NCT03613155
Title: Assessment of Anxiety in Patients Treated by SMUR Toulouse and Receiving MEOPA as Part of Their Care
Acronym: MEOPanx
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/18/0222; 2018-A01687-48 (Other: ID-RCB)
Record Dates: First submitted 2018-07-18; First posted 2018-08-02 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Pain; Anxiety
Keywords: Emergency
MeSH Terms: conditions — Pain; Anxiety Disorders; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Administration of MEOPA as part of the care — Patients should be managed by a SMUR team from Toulouse and benefit from MEOPA administration as part of their management, with a view to analgesia for a painful complaint or prevention of induced pain (for example during mobilization or venous route).

SUMMARY:
The emergency setting, frequently associated with pain and the feeling of loss of control, can cause anxiety in patients.

Reaction anxiety may be an appropriate response to an emergency; Nevertheless, attention must be paid to the evaluation and management of the latter especially as anxiety and pain are closely linked.

DETAILED DESCRIPTION:
There is a definite interest in the management of patients' pre-hospital anxiety. The literature reports a strong association between anxiety, post-traumatic stress and chronic pain. A study conducted at SAMU 31 also found that anxiety on arrival at the emergency department was a negative factor in the treatment of pain. Anxiety can reduce the pain threshold and promote hyperalgesia.

The management of patient anxiety in pre-hospital offers interesting results in terms of analgesia and satisfaction of users of care and should not be neglected.

MEOPA has recently been available in SMUR vehicles (emergency and resuscitation mobile service) at SAMU 31 (urgent medical assistance service); its availability can lead teams to change their practices. More and more emphasis is placed on the importance of positive communication and comfort for which MEOPA, with its conscious sedating effect, could be a facilitating factor.

The aim of our study is to evaluate the level of anxiety of patients treated by SMUR teams in Toulouse and receiving MEOPA following the usual indications for pain-induced pain or pain alleviation.

This is a pilot study, which focuses on the assessment of anxiety in patients treated in pre-hospital care by SMUR Toulouse and receiving MEOPA as part of their care. No data exists in the literature on this subject.

This descriptive study based on qualitative data collected by the FAS1 scale will provide us with the first data on this population. It does not change the usual management of the patient since only patients who must receive MEOPA following the usual indications for pain relief or pain-induced care will be included in the study

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18
* Patient supported by a SMUR team from Toulouse
* Patient receiving MEOPA during pre-hospital care (in the usual indications for pain relief or pain-induced care)
* Patient having given his non-opposition to participate in the study

Exclusion Criteria:

* Any patient with a contraindication to MEOPA:
* Patient requiring pure oxygen ventilation
* Intracranial hypertension
* Any alteration of the state of consciousness preventing the patient's cooperation
* Traumatic brain injury
* Pneumothorax
* Emphysema bubbles
* Gas embolism
* Diving accident
* Abdominal gas distension
* Patient who received an ophthalmic gas for ocular surgery less than three months old
* Known and unsubstituted vitamin B12 deficiency
* Patient under legal protection
* Refusal of the patient to participate in the study
* Barrier of the language or alteration of the communication
* Patient in vital distress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient treated by the SMUR receiving MEOPA during pre-hospital care (in the usual indications for pain relief or pain-induced care)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
The state of anxiety of the patient assessed by Face Anxiety Scale | 2 hours
  The state of anxiety of the patient assessed by FAS (face anxiety scale) self-assessment when supported by a SMUR team with MEOPA administration.
  The FAS, called the Anxiety Faces Scale, is a validated anxiety assessment scale that was originally developed in the context of Critical Care, Critical Care (ICU) management.
  The Faces Anxiety Scale is a valid single-item, self-report measure of state anxiety in intensive care patients that is easy to administer and imposes minimal respondent burden. It has the potential to be a useful instrument for the assessment of state anxiety by clinicians and for research into the reduction of anxiety in this vulnerable population.

SECONDARY OUTCOMES:
The pain felt by the patient, evaluated by the numerical scale (EN), in connection with his anxiety | 2 hours
  EN is a self-rated scale of pain: the patient rates his or her pain on a numeric scale from 0 (no pain) to 10 (maximum pain). The evaluation of the pain at the SAMU is carried out in routine at each support by the EN. For the purposes of this study, the investigators will find the value of the EN in the same temporality as the assessment of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Bounes, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No